CLINICAL TRIAL: NCT05526872
Title: Patient Reminders and Self-Referrals Via Online Patient Portals and Text Messaging (PReVenT) to Improve Adherence to Breast Cancer Screening
Brief Title: A Patient Reminder and Self-Referral Via Online Patient Portals and Text Messaging to Improve Adherence to Breast Cancer Screening
Acronym: PReVenT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Patricia Balthazar, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00004618; NCI-2022-06810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00004618 (Other: Emory University Hospital/Winship Cancer Institute); RAD5676-22 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to their study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (PReVenT intervention) (Experimental): Participants receive usual care as well as a portal message reminder to schedule a SM and a callback link if they need assistance. Participants who have not or do not schedule their SM at the time of the first reminder receive a reminder text-message one week later with a link to receive assistance with scheduling.
  Interventions: Other: Best Practice; Other: Interview; Other: Planned Notification; Other: Survey Administration
- Arm II (enhanced usual care) (Active Comparator): Participants receive usual care as well as portal and text messages one week apart with educational materials about healthy eating.
  Interventions: Other: Best Practice; Behavioral: Health Education; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Behavioral: Health Education — Receive educational materials
  Arms: Arm II (enhanced usual care)
Other: Interview — Ancillary studies
Other: Planned Notification — Receive planned reminders to schedule mammogram
  Other Names: PlannedNotification
  Arms: Arm I (PReVenT intervention)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the patient reminders and self-referrals via online patient portals and text messaging (PReVenT) intervention for improving adherence to breast cancer screening. Though no doctor referral is required for mammography, adherence to screening mammograms remains low. Barriers to screening mammography can include things like forgetfulness, low motivation, high cost, or lack of knowledge. Patient reminders and self-scheduling assistance may overcome some of these barriers by increasing patients' awareness, motivating them to schedule their mammogram, and improving access by removing the need for a healthcare provider to order the exam. The PReVenT intervention uses online and text-message based patient-reminders and self-referral assistance to increase adherence to breast cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES; I. Compare the screening mammogram (SM) completion rates between PReVenT and enhanced usual care (EUC) arms at 6 months.

II. Describe patient's experience with the PReVenT intervention using mixed methods stratified by completion of SM.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive usual care as well as a portal message reminder to schedule a SM and a callback link if they need assistance. Participants who have not or do not schedule their SM at the time of the first reminder receive a reminder text-message one week later with a link to receive assistance with scheduling.

ARM II: Participants receive usual care as well as portal and text messages one week apart with educational materials about healthy eating.

After completion of study, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-74 years
* Active online patient portal account
* Mobile phone number listed in the electronic medical record (EMR)
* At least one primary care visit in our healthcare system between 2015 and 2021
* No screening mammography performed in our healthcare system in the last 2 years

Exclusion Criteria:

* Because of limited research team and patient portal language at this time, non-English speaking patient will be excluded
* Personal history of breast cancer or prior mastectomy
* Participants who already have an upcoming SM scheduled within or outside of Emory Healthcare
* Patients who had a screening mammography at an outside facility within the prior 2 years
* Patients with severe comorbidities at the time of the study (in palliative care or hospitalized at the time of the study)
* Participants who are cognitively impaired or have with history of Alzheimer's disease or dementia

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Completion of Screening Mammogram-Adherence Rate | Within 6 months after enrollment
  Assessed with self-reported surveys and electronic medical record data extraction. Will use chi-square tests and/or two-sample Z-tests for proportions to compare adherence rates between study arms. Fisher's exact test will be considered where necessary.
Completion of Screening Mammogram-Regression Modeling | Within 6 months after enrollment
  Assessed with self-reported surveys and electronic medical record data extraction.Will perform a multivariable logistic regression modeling to compare screening mammogram completion rates between the intervention and control arms while controlling for prior adherence behavior and sociodemographic variables.
Patient Satisfaction-Qualitative | At 6 months
  Will use a mixed-methods approach using surveys and qualitative interviews to evaluate patient satisfaction with the intervention features, online portal and short message service usability i.e., opening the portal message, clicking the embedded link, and replying to the short message service. the patient satisfaction survey measure the following:
  I prefer to get care in person or over the phone instead of using online patient portals, where 1= Strongly Disagree, 2=Disagree, 3= Unsure, 4= Agree, 5= Strongly Agree, 6= Not Applicable. I rarely use online patient portals because I hardly ever need Emory Healthcare services, where 1= Strongly Disagree, 2=Disagree, 3= Unsure, 4= Agree, 5= Strongly Agree, 6= Not Applicable.It was difficult to register for Emory's online patient portal, where 1= Strongly Disagree, 2=Disagree, 3= Unsure, 4= Agree, 5= Strongly Agree, 6= Not Applicable.
Patient Satisfaction-Quantitative | At 6 months
  Will use a mixed-methods approach using chi-square tests and/or two-sample Z-tests for proportions to compare adherence rates between study arms. Fisher's exact test will be considered where necessary.
Assistance with Self-Referral Scheduling | At 6 months
  Will use a mixed-methods approach using surveys and qualitative interviews. Arm I patients will receive a single portal message reminder followed by a single text message reminder with an embedded link to receive a callback to get assistance with self-referral screening mammogram scheduling.The survey measures the following:I only became aware that I was due for screening mammography after I received Emory's online patient portal reminder, where 1= Strongly Disagree, 2=Disagree, 3= Unsure, 4= Agree, 5= Strongly Agree, 6= Not Applicable.I only became aware that I was due for screening mammography after I received Emory's text message reminder, where 1= Strongly Disagree, 2=Disagree, 3= Unsure, 4= Agree, 5= Strongly Agree, 6= Not Applicable.I was more willing to schedule a screening mammography after receiving Emory's online patient portal reminder, where1= Strongly Disagree, 2=Disagree, 3= Unsure, 4= Agree, 5= Strongly Agree, 6= Not Applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Balthazar, MD,CIIP, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT05526872/ICF_000.pdf